CLINICAL TRIAL: NCT04612634
Title: A Randomized, Parallel Controlled Clinical Trial of the Safety and Immunogenicity of Hepatitis A (Live) Vaccine, Freeze-dried in Children Aged 18-24 Months Old
Brief Title: Evaluation of the Safety and Immunogenicity of Hepatitis A Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Changchun Institute of Biological Products Co., Ltd. (Industry); Shaanxi Provincial Center for Disease Control and Prevention (Other); Mianxian Center for Disease Control and Prevention (Unknown); Yangxian Center for Disease Control and Prevention (Unknown); Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JGYM-2020-Ⅳ-01
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Vaccination
MeSH Terms: interventions — Hepatitis A Vaccines; Vaccines; Freeze Drying; Cell Adhesion Molecules

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Research Group 1 (Experimental): 150 subjects are administrated with one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by Changchun Institute of Biological Products Co., Ltd. at the age of 18-24 months old, 0.5 ml each dose, respectively. Blood samples are collected before vaccination and one month (30 days) later.
  Interventions: Biological: Hepatitis A (Live) Vaccine, Freeze-dried produced by Changchun
- Research Group 2 (Active Comparator): 150 subjects are administrated with one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by Zhejiang Pukang Biotechnology Co., Ltd. at the age of 18-24 months old, 0.5 ml each dose, respectively. Blood samples are collected before vaccination and one month (30 days) later.
  Interventions: Biological: Hepatitis A (Live) Vaccine, Freeze-dried produced by Zhejiang
- Research Group 3 (Active Comparator): 150 subjects are administrated with one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. at the age of 18-24 months old, 1.0 ml each dose, respectively. Blood samples are collected before vaccination and one month (30 days) later.
  Interventions: Biological: Hepatitis A (Live) Vaccine, Freeze-dried produced by the Institute of Medical Biology, CAMS

INTERVENTIONS:
Biological: Hepatitis A (Live) Vaccine, Freeze-dried produced by Changchun — Administration of one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by Changchun. 0.5ml per dose
  Arms: Research Group 1
Biological: Hepatitis A (Live) Vaccine, Freeze-dried produced by Zhejiang — Administration of one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by Zhejiang. 0.5ml per dose.
  Arms: Research Group 2
Biological: Hepatitis A (Live) Vaccine, Freeze-dried produced by the Institute of Medical Biology, CAMS — Administration of one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by the Institute of Medical Biology, Chinese Academy of Medical Sciences. 1.0ml per dose.
  Arms: Research Group 3

SUMMARY:
Subjects will be recruited and divided into 3 groups:

1. Hepatitis A（Live）Vaccine，Freeze-dried produced by Changchun Institute of Biological Products Co., Ltd
2. Hepatitis A（Live）Vaccine，Freeze-dried produced by Zhejiang Pukang Biotechnology Co., Ltd., and
3. Hepatitis A（Live）Vaccine，Freeze-dried produced by Institute of Medical Biology, Chinese Academy of Medical Sciences.

After immunization, the immunogenicity and safety of three different manufacturers will be compared and the data will be analyzed.

DETAILED DESCRIPTION:
To evaluate the safety and immunogenicity of Hepatitis A (Live) Vaccine, Freeze-dried produced by Changchhun Institute of Biological Products Co., Ltd, we design this randomized, parallel controlled study. 450 subjects are divided into 3 groups, including 1 experimental group and 2 control groups (Research Group 1, 2, and 3), each group assigned 150 subjects respectively.

All subjects are aged 18-24 months old.

150 subjects from Research Group 1 will be administrated with one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by Changchhun Institute of Biological Products Co., Ltd. Blood samples are collected before vaccination and one month (30 days) later.

150 subjects from Research Group 2 will be administrated with one dose of Hepatitis A（Live）Vaccine，Freeze-dried produced by Zhejiang Pukang Biotechnology Co., Ltd. Blood samples are collected before vaccination and one month (30 days) later.

150 subjects from Research Group 3 will be administrated with one dose of Hepatitis A (Live) Vaccine, Freeze-dried produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. Blood samples are collected before vaccination and one month (30 days) later.

To evaluate the immunogenicity, we will detect and compare the seroconversion rates, and antibody geometric mean concentrations. The safety of all groups will be monitored as well.

ELIGIBILITY:
Inclusion Criteria:

1. subjects aged from 18 to 24 months old at the date of recruitment;
2. with informed consent signed by parent(s) or guardians;
3. parent(s) or guardians are able to attend all planned clinical appointments and obey and follow all study instructions;
4. subjects have not been vaccinated with any type of Hepatitis A vaccines;
5. subjects have no Hepatitis A disease and contraindication of vaccination;
6. subjects did not receive any vaccines within 14 days;
7. before joining this trial, subjects must be qualified and passed their medical history and clinical examinations, and axillary's temperature must be ≤37℃.

Exclusion Criteria:

1. Subjects with history of allergy, convulsion, epilepsy, encephalopathy and psychosis or family history;
2. Allergic to any ingredient of vaccine or with allergy history to any vaccine;
3. Patients with immunodeficiency, in process of cancer treatment, immunosuppressive therapy (oral steroids) or HIV induced hypoimmunity, or in close contact with any family members who has congenital immune diseases;
4. Receive non-specific immunoglobulin within 1 month before recruitment;
5. Subjects with acute febrile diseases with body temperature > 37.0 ℃ or infectious diseases;
6. Subjects with a history of thrombocytopenia or other coagulation disorders that may be contraindicated for hypodermic injection;
7. With known or suspected concurrent diseases include respiratory disease, acute infection or active chronic disease;
8. With severe cardiovascular diseases (Pulmonary heart disease, Pulmonary edema, hypertension cannot be controlled to normal range by drugs), liver and kidney diseases and diabetic complications;
9. Various infectious, suppurative or allergic dermatitis;
10. Other circumstances judged by investigators that are not suitable for this clinical trial.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Antibody Seroconversion rate | 4 months
  Blood samples were collected before and 30 (+ 10) days after immunization. Antibody level and antibody seroconversion rate of HAV-IgG will detect in laboratory. The antibody seroconversion rate of HAV-IgG must maintain the baseline as the other two comparators' products.

SECONDARY OUTCOMES:
Antibody Geometric Mean Titer (GMT) | 4 months
  Antibody GMT will detect in laboratory. The antibody GMT must maintain the baseline as the other two comparators' products.
Adverse Events Incidence rate | 6 months
  Analyse the numbers and rates of participants who suffered from adverse events following immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Shaobai Zhang, Principal Investigator — Shaanxi Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Yangxian Center for Disease Control and Prevention, Hanzhong, Shaanxi
  - Mianxian Center for Disease Control and Prevention, Hanzhong, Shaanxi

IPD SHARING:
Plan to Share IPD: No